CLINICAL TRIAL: NCT05630768
Title: A Multicenter, Open-label, Single-arm Clinical Trial to Evaluate the Efficacy and Safety of Actonel® After Denosumab Discontinuation in Postmenopausal Osteoporosis Women
Brief Title: Efficacy and Safety of Actonel® After Denosumab Discontinuation in Postmenopausal Osteoporosis Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ATN_PMO_IV
Record Dates: First submitted 2022-11-18; First posted 2022-11-30 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2024-12

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Risedronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Actonel® (Experimental): Risedronate Sodium 35mg
  Interventions: Drug: Risedronate Sodium 35 MG [Actonel]; Drug: Calcium Vitamin D combination

INTERVENTIONS:
Drug: Risedronate Sodium 35 MG [Actonel] — Risendronate Sodium Tab. 35mg, orally, once weekly
Drug: Calcium Vitamin D combination — orally, once daily for concomitant drug

SUMMARY:
To evaluate the effect of 1 year of risedronate treatment on the prevention of bone loss after denosumab discontinuation in denosumab-treated post-menopausal osteoporosis for a year

ELIGIBILITY:
Main Inclusion Criteria:

1. Postmenopausal women
2. Patients diagnosed with postmenopausal osteoporosis and administered denosumab for 1 year

Main Exclusion Criteria:

1. Any contraindication to risedronate
2. Those evaluated as inappropriate at the discretion of the investigator

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in lumbar spine bone mineral density (LS BMD) at 1 year (%) | 1 year
  Percent change from baseline in lumbar spine bone mineral density (LS BMD) at 1 year (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seodaemun-gu, South Korea